CLINICAL TRIAL: NCT00868803
Title: Identification of Aberant Gene Expression in Human Prostatic Carcinoma
Brief Title: Aberrant Gene Expression Prostate Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Linda Topjian, study coordinator, Lahey Clinic
Other Study IDs: LCID1995-014
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surplus tissue following pathologic review requirements will be snap frozen and processed for extraction of RNA. mRNA will be reversed transcribed to make cDNA with the prime 5'TCCTTAGAAC, followed by 40 cycles of palindromic PCR using the sam eprimer. Amplified cDNA (35 S-labled) will be analysed on a 4% polyacrylamide gel. Comparative analysis of cDNA amplified products will serve to identify aberrantly expressed candidate genes. Such products will be isolated, sequenced and evaluated as to their role in establishing the neoplastic pheotype and the potential utility as a marker of prostatic neoplastic progression.
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is to gain a better understanding of the molecular changes responsible for causing prostate cancer and that examination of tissue and blood samples will help in the development of improved screening and therapeutic approaches.

DETAILED DESCRIPTION:
The goal of this study is to identify novel genetic elements that are aberantly expressed throughout prostatic neoplastic progression. The approaches proposed exploit the known familial arm of prostatic cancer, using established molecular genetic approaches, and extend these studies to sporadic prostatic cancer using a novel technique of differential display. Application of the latter technique to colon cancer in the American population establishes this tumor type as a high priority for scientific investigation and this study is part of an initiative to address this problem. Presently the studies in the field of prostate are under-represented. The collection of tissue samples from patients diagnosed with prostate cancer. Patients will also provide a blood sample at the time of their surgery and potentially post-op from 6 mos to 5 years. Samples will also be obtained from patients who's biopsy turns out to be non-prostate cancer. These samples will be obtained shortly following the biopsy out to 6 months after the biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed prostate cancer undergoing prostatectomy
* Suspicion of prostate cancer undergoing biopsy - negative biopsy
* Health volunteer (control group) - blood sample for PSA

Exclusion Criteria:

* Patients not fitting the inclusion criteria

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with prostate cancer patients undergoing surgery for suspected prostate cancer but have negative biopsy healthy volunteers - blood sample only
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1995-04; Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly R Christ, PhD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States